CLINICAL TRIAL: NCT04495062
Title: Acquisition of Physiological Signals With a Wearable Technology to Assist on Research Aiming to Improve Early Identification of Exacerbations in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: The Use of Wearable Technology to Acquire Signals for COPD Research
Status: Completed | Type: Observational
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other); Acurable Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 19/NI/0194
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a respiratory condition which affects approximately 3 million people in the UK and 210 million worldwide. The disease is characterized by progressive air flow obstruction and decline of lung function. COPD is currently the fourth leading cause of death in the world. The main reason for hospitalisations associated with COPD is exacerbations (chest infections or a worsening of the underlying symptoms). Severe COPD exacerbations are the second largest cause of emergency admissions in the UK. Mild and moderate exacerbations can be managed in the community but if they are not identified promptly they may progress to breathlessness and in some patients to respiratory failure. Thus, finding modalities for early detection and diagnosis of exacerbations is clearly a priority for current and future COPD research. However, these still do not exist. The aim of this study will be to acquire acoustic respiratory signals from COPD patients with a small wearable device. These signals will be subsequently used to carry out engineering research with the objective of trying to find "fingerprints" in them which could be early indicators of disease exacerbations. If those "fingerprints" were found, subsequent research could focus on trying to create software methods which, together with the use of a small wearable device, would aim at automatically detecting exacerbations when they are at very early stages- prior to the symptoms being evident to the patient- so that clinical intervention could be triggered, in order to optimize the disease outcomes.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a condition characterised by progressive air-flow obstruction, decline in lung function caused by airway inflammation and damaging of air sacs. The resulting narrowing of airways makes it harder to breathe in and out. COPD is currently the fourth leading cause of death worldwide and in the UK the National Institute for Health and Clinical Excellence (NICE) estimates that the total direct cost of COPD to the NHS is over £800million - out of which £300 million correspond to hospitalisations.

Therefore, it is widely acknowledged that anything that improves management and effectiveness of treatment will not only improve patients' quality of life but also result in savings from: 1) Emergency hospital admissions; 2) Potential GP visit; 3) Loss of productivity due to work in absenteeism.

Severe COPD exacerbations (periods where there is acute worsening of respiratory symptoms such as cough, dyspnoea, wheezing, increased sputum production) cause one in eight hospital admissions. Mild and moderate exacerbations can be managed outside hospital but if not identified and treated promptly may progress in some patients to respiratory failure. A significant proportion of these exacerbations will require inpatient treatment and can reduce the quality of life of patients increasing their morbidity and mortality. Thus, finding modalities for early detection and diagnosis of exacerbations is clearly a priority in current and future COPD research, but currently these still do no exist.

The longer term goal of our research is to have a novel acoustic based wearable wireless technology that will be able to monitor COPD patients for extended periods of time, and automatically provide early detection of potential exacerbations even prior to symptoms which can be treated promptly to minimise their likelihood of progression to higher levels of severity.

We have developed a small wearable device which is easy to use and for the first time allows continuous non-intrusive recordings of respiratory sounds and more specifically has been designed to optimise transmission of the acoustic signals generated by airflow within the trachea.

We will aim to acquire signals from two groups of COPD patients:

1. A group undergoing exacerbations
2. A second group of stable, potential exacerbators, COPD patients

The group of patients undergoing exacerbations will be recruited from medical wards and patients who agree to participate in the trial will be fitted with the device during their inpatient stay. Clinical data will be collected including but not limited to: co-morbidities, medications, oxygen given; timing of exacerbations medications (antibiotics, steroids, nebulisers) and observations. Patients will also be given a diary to complete during their inpatient stay for when they are ambulating, documentation of sputum production as well as other activities. Patients will also be given the option of taking the device home for several days whilst recovering from their exacerbation.

The stable patients will be recruited from outpatient clinics and if clinically stable trained to use a device to take home for a pre-agreed period of time, up to one month. They will be expected to wear the device at night whilst sleeping and will have support throughout if needed. They will also be asked to complete a diary which documents amongst other things, sputum production, any exacerbations, symptoms, exercise and a range of other activities.

Patients in both groups will be given usability questionnaires regarding comfort, usability, ease of the device and also be invited to attend focus groups to feedback about the device.

The study will aim to develop a novel acoustic based wearable technology which will in the long term monitor COPD patients for an extended time period and automatically provide early detection of potential exacerbations. This has several benefits including:

1. Disease management optimisation resulting in better quality of life and lower severity of symptoms
2. Prompt and early treatment of exacerbations leading to fewer hospital admissions and can slow disease progression
3. Can potentially result in more personalised treatment and management, with efficient use of drugs and reduction in treatment cost.

ELIGIBILITY:
Inclusion criteria:

• Patients with a diagnosis of COPD (FEV1:FVC <0.7)

Exclusion Criteria:

* Age < 18 or >80years
* Subjects who are not fluent in English, or who have special communication needs.
* Known allergy to the adhesive dressing.
* For the stable patients, subjects with physical or mental impairments who would not be able to use the new technology on their own.
* Subjects with very loose/saggy skin in the neck area which would unavoidably result in the device swinging if moving the neck.
* Subjects with implantable devices
* Subjects with known sleep disordered breathing
* Subjects with stridor
* Subjects requiring ventilation
* Subjects unable to give consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a proven diagnosis of chronic obstructive pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
The primary objective of this work is to acquire acoustic signals from two groups of COPD patients, that can subsequently be used to carry out COPD signal processing research. | Signals will be recorded for a maximum of 4 weeks
  Acoustic signals from wearable technology will be collected from stable COPD patients but also patients with an exacerbation of COPD and the signals analysed for changes

SECONDARY OUTCOMES:
To explore the usability aspects of a small wearable device in the context of COPD patients | 2 patient visits lasting a maximum 1 hour.
  Usability questionnaires and patient focus and feedback groups will be used to get feedback about the device

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Respiratory Department Royal Free Hospital NHS Foundation Trust, London, United Kingdom